CLINICAL TRIAL: NCT07128433
Title: Prospective Randomized Controlled Clinical Trial on the Impact of Antepartum Breast Milk Expression on Breastfeeding Rates in Patients With Gestational Diabetes Mellitus
Brief Title: Impact of Antepartum Breast Milk Expression on Breastfeeding Rates in Patients With Gestational Diabetes Mellitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025R0084-0001
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Gestatiaonl Diabetes Mellitus
Keywords: Antepartum; milk expression; Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antepartum Milk Expression Group (Active Comparator): Oarticipants will receive one-on-one antenatal breast milk expression instruction by a midwife and initiate twice-daily practice from 37 weeks gestation onward.
  Interventions: Procedure: milk expression
- Control group (No Intervention): Participants will receive routine antenatal care and standard postpartum management

INTERVENTIONS:
Procedure: milk expression — Following one-on-one antenatal manual colostrum expression instruction by a midwife at the breastfeeding clinic, participants will initiate twice-daily practice from 37 weeks gestation onward, performing 3-5 minutes of manual expression per breast per session (total duration ≤10 minutes per session).
  Arms: Antepartum Milk Expression Group

SUMMARY:
This study proposes a prospective randomized controlled clinical trial involving primiparous women diagnosed with gestational diabetes mellitus (GDM) carrying singleton pregnancies. Participants will be randomized in a 1:1 ratio into either a control group or an intervention group.

The control group will receive standard prenatal care followed by routine postpartum breastfeeding guidance.

In addition to the standard care provided to the control group, the intervention group will receive one-on-one midwife-led manual breast milk expression training at the breastfeeding clinic. They will begin manual expression twice daily starting at 37 weeks gestation.

The primary outcome will compare exclusive breastfeeding rates at 3 months postpartum between groups through postpartum follow-up assessments to evaluate the impact of antenatal milk expression on breastfeeding success in GDM patients.

ELIGIBILITY:
Inclusion Criteria:

* Expressed intention for exclusive breastfeeding; Aged 20-45 years; Nulliparous status; Singleton pregnancy; GDM diagnosed per 75g OGTT at 24-28 weeks

Exclusion Criteria:

* Contraindications to breastfeeding; multifetal pregnancy; placenta previa; pregestational diabetes mellitus; preeclampsia; contraindications to vaginal delivery; fetal structural anomalies (cleft lip/palate, cardiac malformations, neural tube defects); chromosomal abnormalities or metabolic disorders affecting suckling ability (e.g., phenylketonuria); intrauterine growth restriction; macrosomia; polyhydramnios; maternal psychiatric disorders (depression or anxiety disorders)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Biologically female individuals capable of conception and childbirth
Enrollment: 212 (Estimated)
Dates: Start 2025-08-19 (Estimated); Primary Completion 2027-08-18 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Exclusive breastfeeding rates at 3 months postpartum | 3 months postpartum

IPD SHARING:
Plan to Share IPD: Undecided